CLINICAL TRIAL: NCT01753583
Title: High-resolution Imaging of Corneal Lesions With Optical Coherence Tomography (OCT) - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-041112
Record Dates: First submitted 2012-12-07; First posted 2012-12-20 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Corneal Abrasions; Corneal Infiltrates
Keywords: optical coherence tomography; corneal abrasion; corneal infiltrate
MeSH Terms: conditions — Corneal Injuries | interventions — Tomography, Optical Coherence; Slit Lamp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 patients with corneal abrasions (Experimental)
  Interventions: Device: Optical Coherence Tomography (OCT); Other: Slit lamp biomicroscopy
- 10 patients with corneal infiltrates (Experimental)
  Interventions: Device: Optical Coherence Tomography (OCT); Other: Slit lamp biomicroscopy

INTERVENTIONS:
Device: Optical Coherence Tomography (OCT) — High-resolution OCT imaging of the cornea
Other: Slit lamp biomicroscopy — Slit lamp biomicroscopy with fluorescein staining and slit lamp photograph

SUMMARY:
Corneal lesions such as corneal abrasions and corneal infiltrates are common in clinical practice. The current study seeks to investigate whether high-resolution OCT is suitable for imaging of these corneal lesions. The present study has the character of a pilot study and the results are intended to be used to develop a standardized protocol for imaging and analysis of these corneal lesions. Based on this protocol, further studies investigating the pathophysiology of corneal lesions or evaluating therapeutic success can be planned.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Newly diagnosed corneal abrasion or corneal infiltrate

Exclusion Criteria:

* Recurrent corneal erosion
* Participation in a clinical trial in the previous 3 weeks
* Presence of any abnormalities preventing reliable measurements as judged by the investigator
* Any contraindication for topical application of Novain 0.4% eye drops for topical anesthesia or of Minims-Fluorescein Sodium eye drops for fluorescein staining
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Imaging of corneal abrasions and infiltrates | 1 day
  The aim of this pilot study is to investigate whether imaging of these corneal alterations is possible.

SECONDARY OUTCOMES:
Size and depth of corneal lesions as assessed with high-resolution OCT | 1 day
  The volume and size of corneal lesions or infiltrates will be assessed using a specific software.
Slit lamp biomicroscopy with fluorescein staining | 1 day
  The volume and size of corneal lesions or infiltrates will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria